CLINICAL TRIAL: NCT06531590
Title: Emergency Department Management of Anterior Shoulder Dislocation Patients
Brief Title: Anterior Shoulder Dislocation at Emergency Department
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Ankara Etlik City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: anterior shoulder dislocation
Record Dates: First submitted 2024-07-17; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Shoulder Dislocation; Analgesia; Pain, Shoulder
Keywords: shoulder dislocation; interscalene nerve block; suprascapular nerve block; intraarticular lidocaine injection; emergency department
MeSH Terms: conditions — Shoulder Dislocation; Agnosia; Shoulder Pain; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ketamine group: patients receiving ketamine as analgesic after shoulder dislocation
- intraarticular lidocaine injection group: patients receiving intraarticular lidocaine injection as analgesic after shoulder dislocation
- interscalene nerve block group: patients receiving interscalene nerve block group as analgesic after shoulder dislocation
- suprascapular nerve block group: patients receiving suprascapular nerve block group as analgesic after shoulder dislocation

SUMMARY:
In this study, investigator will analyze the demographic characteristics of patients presenting to emergency department with Anterior Shoulder Dislocation. Investigators will document the mechanism of injury, orthopedic classification of shoulder dislocation, associated treatments, pre-procedural pain scoring, post-procedural pain scoring, as well as the duration of emergency department stay related to the preferred treatment, orthopedic consultation, and patient outcomes (discharge, admission to ward or intensive care unit, mortality). Aim of the study to investigate whether the current treatments used provide any superiority in emergency department outcomes for patients

DETAILED DESCRIPTION:
Intravenous analgesia (Paracetamol, NSAIDs, opioids) is preferred for patients during the treatment and reduction stages of anterior shoulder dislocation. Additionally, patients may receive regional anesthesia and analgesia (lidocaine, bupivacaine). The route and dosage of analgesic administration are chosen by the attending physician managing the patient. In this study, investigators plan to observationally evaluate the analgesic management of patients without intervening in the method and dosage chosen by the primary treating physician.

Patients receiving analgesia will be chosen according to preffered treatment at emergency department. The study population will consist of patients presenting to the emergency department with shoulder dislocation who receive analgesia and fall into the following 4 treatment groups.

These 4 group will consist in:

1. ketamine group
2. interscalene nerve block group
3. suprascapular nerve block group
4. intraarticular lidocaine injection group. The study will compare these 4 treatment methods in terms of analgesia management, reduction time, comfort, and length of hospital stay for patients presenting to the emergency department with shoulder dislocation and receiving analgesia. The researcher will not interfere with the treatment decision made by the responsible physician or the treatment process

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years and older

Exclusion Criteria:

Patients who are not conscious at the time of admission and do not consent to participate in the study.

Patients who do not have follow-up in our healthcare system or cannot be followed up.

Patients with allergies to opioids or local anesthetics. Patients presenting to the emergency department with suspicion of multiple fractures and dislocations involving ≥2 different types of injuries will also be excluded from the study.

Forensic cases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients followed at emergency department after shoulder dislocation who received analgesic treatment
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
shoulder reduction | 24 hours
  succesful reduction of shoulder joint and assessment of pain before and after analgesic treatments with pain scales ( visual analogue scale, verbal pain intensity scale, PAINAD ( pain assessment in advanced dementia) scale andvisual analogue scale)

CONTACTS AND LOCATIONS:
Overall Officials: gulsen akcay, ass. prof., Study Director — ass. prof. of organization
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buren MA, Theologis A, Zuraek A, Behrends M, Clark AJ, Leung JM. Lidocaine Infusion for the Management of Postoperative Pain and Delirium (LIMPP): protocol for a randomised control trial. BMJ Open. 2022 Jun 6;12(6):e059416. doi: 10.1136/bmjopen-2021-059416. PMID 35667730
- [Background] Hayashi M, Kano K, Kuroda N, Yamamoto N, Shiroshita A, Kataoka Y. Comparative efficacy of sedation or analgesia methods for reduction of anterior shoulder dislocation: A systematic review and network meta-analysis. Acad Emerg Med. 2022 Oct;29(10):1160-1171. doi: 10.1111/acem.14568. Epub 2022 Aug 11. PMID 35872652
- [Background] Gawel RJ, Grill R, Bradley N, Luong J, Au AK. Ultrasound-Guided Peripheral Nerve Blocks for Shoulder Dislocation in the Emergency Department: A Systemic Review. J Emerg Med. 2023 Nov;65(5):e403-e413. doi: 10.1016/j.jemermed.2023.05.021. Epub 2023 Jun 9. PMID 37741738